CLINICAL TRIAL: NCT05447091
Title: Examining the Effectiveness of a Custom-made Tablet-based Video Game Intervention on Mood and Cognition in Adults
Brief Title: Examining the Effectiveness of a Tablet Video Game on Mood and Cognition
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: aMoon fund (Unknown)
Responsible Party: Principal Investigator, Mor Nahum, Principal Investigator, Hebrew University of Jerusalem
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Thrive
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Mood Disturbance; Depressive Symptoms
Keywords: Cognitove Control; Video-games; Cognitive Control Training
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are not aware of the treatment group they are assigned to. The PI is not aware of the treatment condition in which participants are. Finally, the assessors are blinded to the group assignment as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active high dose treatment (Active Comparator): Active LOH game training- high dose
  Interventions: Behavioral: LOH game- high dose
- Active low dose treatment (Active Comparator): Acrive LOH game training - low dose
  Interventions: Behavioral: LOH game- low dose
- Sham treatment (Sham Comparator): Sham LOH game- high dose
  Interventions: Behavioral: LOH sham game

INTERVENTIONS:
Behavioral: LOH game- high dose — Participants will be asked to complete 15 half-hour training sessions, over 3 weeks, ie about 5 training sessions a week, and a total of 7.5 hours of training for 3 weeks.
  Arms: Active high dose treatment
Behavioral: LOH game- low dose — Participants will be asked to complete 6 half-hour training sessions, over 3 weeks, ie about 2 training sessions a week, and a total of 3 hours of training for 3 weeks.
  Arms: Active low dose treatment
Behavioral: LOH sham game — Participants will be asked to complete 15 half-hour training sessions, over three weeks, using sham version of the game. the sham version does not include components of cognitive training.
  Arms: Sham treatment

SUMMARY:
Sustained negative mood and depression are characterized by functional impairment, and significant reduction in quality of life. Cognitive models of depression emphasize the role of impaired cognitive control - the mental abilities determining goal directed behaviors - in contributing to depressive symptoms. Indeed, research findings from subclinical and clinical populations show that depressive symptoms are associated with decreased cognitive control abilities.

The THRIVE trial is a double-blind, proof-of-concept randomized controlled trial (RCT). The aims of the study are to investigate the feasibility and efficacy of an innovative, custom-made tablet video game, Legends of Hoa'manu (LOH), which is designed to enhance cognitive control, in alleviating mood and improving cognitive control in adults.

Participants with mild to major depressive symptoms will be randomized to receive either LoH or a control intervention. Cognitive control, mood and depressive symptoms will be assessed at baseline, post training, after at a 3-week and a 3-month follow up.

DETAILED DESCRIPTION:
Persistent negative mood, melancholy and depression are becoming more and more prevalent worldwide. Depression is linked to severe functional impairment, which can last for years, and to a significant reduction in quality of life. Current theoretical models of depression suggest that negative mood and depressive symptoms are associated with decreases in cognitive control abilities - the same brain mechanisms in the prefrontal cortex that underlie goal-directed behaviors. Specifically, difficulty in delaying a response to irrelevant negative information, or difficulty in removing irrelevant negative information from working memory, have all been found to be associated with and predictive of depressive symptoms. Indeed, research findings from subclinical and clinical populations show that depressive symptoms are associated with decreased cognitive control ability and decreased activity in the prefrontal cortex regions.

In the present study, the investigators will examine whether training of cognitive control improves mood. Specifically, the investigators will test whether several weeks of training using a tablet video game targeting cognitive control improves depressive symptoms, mood, and cognitive control abilities measures among adults. Participants will be randomized to receive either a high or low dose of the intervention or a control intervention, and will be asked to train with their intervention remotely from home for 3 weeks. Outcomes will be assessed at baseline, at the completion of training and at two follow up points: 3 weeks and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and woman 18-60 years of age.
* Symptoms at a minimal level and above of depression, according to a score of 5 or higher in the Personal Health Questionnaire Depression Scale (PHQ-8).
* Able and interested in signing an informed consent form.
* speak and read Hebrew, English or Russian.

Exclusion Criteria:

* Video game addiction disorder.
* Neurological diseases that cause cognitive decline (such as dementia), based on self-report.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI-II) | 3 weeks
  To assess levels and change of depressive symptoms. The BDI-II consists of 21-items, scored on a Likert scale from 0 to 3 (range 0-63), and has demonstrated high reliability and good concurrent, content, and structural validity for screening depression in outpatient and student samples.

SECONDARY OUTCOMES:
Ruminative Responses Scale-Short Version (RRS-10) | 3 weeks
  To assess level and change of ruminative responses. It is a 10-item self-report measure with a 4-point Likert scale (1=almost never; 4=almostalways) comprised of two subscales: Brooding (e.g., 'Think "Why do I always react thisway?"'; 'Think "Why do I have problems other people don't have?"') and Reflection (e.g.,'Write down what you are thinking and analyze it'; 'Go someplace alone to think aboutyour feelings'). Scores for each subscale are computed by summing its respective items.Higher scores indicate higher rumination levels. The internal consistency values observedin the original study werea=.77 anda=.72 for Brooding and Reflection subscales.
Generalised Anxiety Disorder-7 (GAD7) | 3 weeks
  To assess level and change of anxiety symptoms. It is a self-rated, validated screening instrument for anxiety and measures its severity. It has 7 items which are evaluated as 0 being not at all, to 3, nearly every day. Based on the total score of the individual, anxiety is categorised as none (0-4), mild (5-9), moderate (10-14), and severe (15-21) reflecting the degree of anxiety.
Adaptive Cognitive Evaluation (ACE) | 3 weeks
  To assess level and change of cognitive control. The ACE is a mobile assessment battery containing standard tests that assess different aspects of cognitive control (attention, working memory, and goal management).
WHO-5 Well-Being Index (WHO-5) | 3 weeks
  To assess level and change of well-being. The WHO-5 is a short, self-administered measure of well-being over the last two weeks. It consists of five positively worded items that are rated on 6-point Likert scale, ranging from 0 (at no the time) to 5 (all of the time). The raw scores are transformed to a score from 0 to 100, with lower scores indicating worse well-being. A score of ≤50 indicates poor wellbeing and suggests further investigation into possible symptoms of depression. A score of 28 or below is indicative of depression.

OTHER OUTCOMES:
Satisfaction with the intervention questionnaire | 3 weeks
  It is a 20-item self-report questionnaire with a 7-point Likert scale (1=Do not agree at all; 4=Agree most)

CONTACTS AND LOCATIONS:
Overall Officials: Mor Nahum, PhD, Principal Investigator — Hebrew University of Jerusalem
Locations (1):
- Computerized Neurotherapy Lab, School of OT, Hebrew University, Mt. Scopus Campus, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No